CLINICAL TRIAL: NCT03868579
Title: A Pilot Study to Evaluate the Diagnostic Performance of Pleural Touch Preparations in Pleuroscopy, a Prospective Study
Brief Title: Rapid On Site Evaluation of Pleural Touch Preparations in Diagnosing Malignant Pleural Effusion in Patients Undergoing Pleuroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-0746; NCI-2019-00735 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0746 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-03-07; First posted 2019-03-11 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Malignant Neoplasm; Malignant Respiratory Tract Neoplasm; Malignant Thoracic Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Biopsy; Thoracoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observational (pleuroscopy, medical chart review) (Experimental): Patients undergo biopsy of the lining of the lung using pleuroscopy. Medical chart of patients is also reviewed.
  Interventions: Procedure: Biopsy; Other: Medical Chart Review; Procedure: Thoracoscopy

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: Bx
Other: Medical Chart Review — Review medical chart
  Other Names: Chart Review
Procedure: Thoracoscopy — Undergo pleuroscopy

SUMMARY:
This trial studies how well rapid on site evaluation of pleural touch preparations works in diagnosing cancerous fluid in between the linings of the lungs (malignant pleural effusion) in patients undergoing a pleuroscopy. A type of laboratory testing called rapid on site evaluation of pleural touch preparations that uses pleural biopsy tissue samples collected during an already-scheduled pleuroscopy may be able to diagnose malignant pleural effusion.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the specificity of rapid on site evaluation (ROSE) of touch preparations (preps) for predicting malignancy on final pathology in pleuroscopy.

SECONDARY OBJECTIVES:

I. To estimate the sensitivity of rapid on site evaluation (ROSE) of touch preparations (preps) for predicting malignancy on final pathology in pleuroscopy.

II. To estimate the specificity and sensitivity of visual assessment of pleura for predicting malignancy on final pathology in pleuroscopy.

III. To compare the specificity and sensitivity of ROSE of touch preps between centers.

OUTLINE:

Patients undergo biopsy of the lining of the lung using pleuroscopy. Medical chart of patients is also reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo pleuroscopy with biopsy

Exclusion Criteria:

* Patients with known malignant pleural effusion
* Inability or unwillingness to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Specificity of rapid on site evaluation (ROSE) of touch preparations (preps) for predicting malignancy | Up to 1 year
  Descriptive statistics (e.g., frequencies, ranges, means, medians, proportions, and standard deviations [SDs]) along with 95% confidence intervals (CIs) for the means or proportions will be computed for the measures of interest. Specificity will be defined as true negative (TN) divided by (TN + false positive [FP]). High probability of malignancy is defined as adequate tissue with tumor present. Low probability of malignancy defined is adequate tissue with no tumor present. Indeterminate probability of malignancy is defined as presence of atypical cells but inadequate for a definitive diagnosis on ROSE. Will collapse the indeterminate probability of malignancy (atypical cells category) found on touch preps into low probability for malignancy bin and indeterminate probability of malignancy on visual assessment into low probability for malignancy.

SECONDARY OUTCOMES:
Sensitivity of ROSE of preps for predicting malignancy | Up to 1 year
  Descriptive statistics (e.g., frequencies, ranges, means, medians, proportions, and SDs) along with 95% CIs for the means or proportions will be computed for the measures of interest. Sensitivity will be defined as true positive (TP) divided by (TP + false negative [FN]). High probability of malignancy is defined as adequate tissue with tumor present. Low probability of malignancy defined is adequate tissue with no tumor present. Indeterminate probability of malignancy is defined as presence of atypical cells but inadequate for a definitive diagnosis on ROSE. Will collapse the indeterminate probability of malignancy (atypical cells category) found on touch preps into low probability for malignancy bin and indeterminate probability of malignancy on visual assessment into low probability for malignancy.
Specificity of visual assessment of pleura for predicting malignancy | Up to 1 year
  Descriptive statistics (e.g., frequencies, ranges, means, medians, proportions, and SDs) along with 95% CIs for the means or proportions will be computed for the measures of interest. Specificity will be defined as TN divided by (TN + FP). High probability of malignancy is defined as presence of abnormalities, such as studding, presence of parietal or visceral masses or nodules, or abnormal tissue deposits consistent with malignancy. Low probability is defined as absence of abnormalities or presence of purulent, fibrino-purulent pleural fluid or parietal and/or visceral pleura inflammation or thickening. Indeterminate probability is defined as findings which cannot include or exclude malignancy with certainty, such as inflammation of the pleura or adhesions, but that cannot be classified by the interventionist in any of the above categories. Will collapse the indeterminate probability of malignancy on visual assessment into low probability for malignancy.
Sensitivity of visual assessment of pleura for predicting malignancy | Up to 1 year
  Descriptive statistics (e.g., frequencies, ranges, means, medians, proportions, and SDs) along with 95% CIs for the means or proportions will be computed for the measures of interest. Sensitivity will be defined as TP divided by (TP + FN). High probability of malignancy is defined as presence of abnormalities, such as studding, presence of parietal or visceral masses or nodules, or abnormal tissue deposits consistent with malignancy. Low probability is defined as absence of abnormalities or presence of purulent, fibrino-purulent pleural fluid or parietal and/or visceral pleura inflammation or thickening. Indeterminate probability is defined as findings which cannot include or exclude malignancy with certainty, such as inflammation of the pleura or adhesions, but that cannot be classified by the interventionist in any of the above categories. Will collapse the indeterminate probability of malignancy on visual assessment into low probability for malignancy.
Positive predictive value (PPV) for all patients | Up to 1 year
  PPV will be defined as TP divided by (TP + FP). Pre-test odds will be calculated using the formula: pre-test probability divided by (1 - pre-test probability). Post-test odds will be calculated using the formula: pre-test odds times likelihood ratio, and post-test probability was calculated using the formula: post-test odds divided by (1 + post-test odds). Likelihood ratios (LRs) will also be calculated by dividing the probability of a result in patients with the disease by the probability of the same result in patients without the disease.
Negative predictive value (NPV) for all patients | Up to 1 year
  NPV will be defined as TN divided by (TN + FN). Pre-test odds will be calculated using the formula: pre-test probability divided by (1 - pre-test probability). Post-test odds will be calculated using the formula: pre-test odds times likelihood ratio, and post-test probability was calculated using the formula: post-test odds divided by (1 + post-test odds). LRs will also be calculated by dividing the probability of a result in patients with the disease by the probability of the same result in patients without the disease.
Specificity of ROSE on touch preps between centers | Up to 1 year
  Will be compared between centers using Chi-squared and Fisher exact tests.
Sensitivity of ROSE on touch preps between centers | Up to 1 year
  Will be compared between centers using Chi-squared and Fisher exact tests.

CONTACTS AND LOCATIONS:
Overall Officials: Horiana Grosu, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (3):
  - Mayo Clinic, Rochester, Minnesota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
- Nicosia General Hospital, Nicosia, Cyprus

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT03868579/ICF_000.pdf